CLINICAL TRIAL: NCT03334123
Title: Effects of Exercise and Exercise Counselling in Hemodialysis Patients: a Randomized Controlled Trial.
Brief Title: Effects of Exercise and Exercise Counselling in Hemodialysis Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Jernej Pajek, Jernej Pajek, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DIAGIBII
Record Dates: First submitted 2017-10-10; First posted 2017-11-07 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Physical Activity; Kidney Diseases; Kidney Failure; Chronic Kidney Diseases; End Stage Renal Disease
Keywords: exercise; aerobic exercise; functional training; strength training; resistance training; kidney failure; rehabilitation; physical activity; hemodialysis; dialysis patients; chronic renal failure; chronic kidney disease; end-stage renal disease; intradialytic exercise
MeSH Terms: conditions — Motor Activity; Kidney Diseases; Renal Insufficiency; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional training and cycling (Experimental): Participants in this group will perform 20 minutes of functional training before dialysis (in the first 8 weeks) and intradialysis cycling exercise during dialysis. Participants will also receive exercise counselling; investigators will teach them how to practice at home by practice and examples given during the 20 minutes of functional training pre-dialysis. In the second phase of additional eight weeks participants will perform the functional training at home on non-dialysis days in addition to intradialysis cycling. Kinesiologist will monitor, advice and motivate them.
  Interventions: Other: Functional training and cycling
- Cycling (Active Comparator): This active control comparator group will perform intradialytic cycling on an adapted ergometer 3 times per week for 4 months without functional training prior to dialysis procedure and without exercise counselling.
  Interventions: Other: Cycling

INTERVENTIONS:
Other: Functional training and cycling — First 8 weeks: patients will perform 20 minutes of functional training before their dialysis procedure. The exercise program will be run by kinesiologists, who will also teach patients how to perform exercises on their own at home. During intradialysis cycling 3 times weekly participants will cycle on adapted ergometer. Participants will start with 10 - 15 minutes of cycling and then gradually increase time and intensity up to 45 minutes of duration.
  Second phase of 8 weeks: participants will no longer perform functional training before dialysis but will be motivated, monitored and advised to perform functional exercise at home on non-dialysis days for 20-30 minutes and continue with cycling sessions during the dialysis procedures three times weekly.
  Other Names: Functional training, intradialysis cycling and counselling; Experimental group
  Arms: Functional training and cycling
Other: Cycling — First 8 weeks: cycling on an adapted ergometer during dialysis; starting with 10 - 15 minutes of cycling and then gradually increasing time and intensity up to 45 minutes of duration.
  Second 8 weeks: continue with cycling at the target duration and intensity during dialysis.
  Other Names: Intradialysis cycling exercise; Active control group
  Arms: Cycling

SUMMARY:
The aim of the study is to determine the effect of functional exercise and training counseling by kinesiotherapist in addition to the basic exercise program of cycling during dialysis on physical performance of dialysis patients.

DETAILED DESCRIPTION:
Study will include 86 dialysis patients. Investigators will first test the strength of lower limbs with sit-to-stand test, handgrip strength, flexibility, balance, submaximal aerobic capacity, physical characteristics and clinical parameters. After that randomization of patients in two groups will be made - one experimental and one active control group. Patients who will refuse to exercise will be invited to a non-randomized inactive control group (without exercise).

The experimental group will attend 3 times weekly a guided functional exercise before the dialysis procedure for 20 minutes and perform a cycling session during dialysis in the first phase of the study, which will last for 8 weeks. During this time experimental group will receive exercise counselling; instructions how to practice at home will be given by examples and training during functional exercise predialysis sessions.

In the second phase of the study for additional eight weeks participants will be instructed to exercise at home using the skills mastered during the first study phase on non-dialysis days, and continue with the program of intradialysis cycling. Investigators will give them advice, monitor and motivate them.

The active control group will perform intradialytic exercise (intradialysis cycling equal to cycling program of experimental group) during dialysis procedure for four months.

The primary end-point of the study is a change in the 10-repetition sit-to-stand test time as a measure of strength of lower extremities.

Exercise program will be run by a kinesiologist. Main hypothesis is that the guided functional exercise under the surveillance of a kinesiologist added to intradialysis cycling program statistically significantly improves patient's physical performance as compared to the program of intradialysis cycling alone.

ELIGIBILITY:
Inclusion Criteria:

* dialysis patients on renal replacement therapy with chronic hemodialysis,
* duration of hemodialysis treatment for at least 3 months,
* age 18-90 years,
* capable of independent walking and independent feeding.

Exclusion Criteria:

* the presence of chronic malignant or infectious disease,
* uncontrolled arterial hypertension with an average of the last five pre-dialysis blood pressure values above 180/100 mm Hg,
* unstable angina pectoris or Canadian Cardiovascular Society class 2-4,
* heart failure New York Heart Association class 3 and 4,
* the presence of a psychotic illness or a mental disability,
* a condition with an amputated limb (more than 2 fingers on the lower limb and / or more than 2 fingers on the upper limb)
* any other condition that causes the clinical unstability of the patient (i.e. repetitive gastrointestinal hemmorrhagies, liver cirrhosis with frequent exacerbations, advanced dementia with poor cooperation of the patient)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in 10 repetition sit-to-stand test time | baseline, 8 weeks and 16 weeks
  Performance of the sit-to-stand test involves activation of the lower limb muscles; the test measures lower limb strength. Participants are required to 10 times stand up from and sit down on an armless chair as quickly as possible. Their arms should be folded across their chest.

SECONDARY OUTCOMES:
Change in 6-minute walk test distance | baseline, 8 weeks and 16 weeks
  Distance made in 6-minute walk test (submaximal aerobic endurance)
Change in lean and fat body mass | baseline, 8 weeks and 16 weeks
  Body composition measurements by bioimpedance
Change in serum interleukin-6 (IL-6) | baseline, 8 weeks and 16 weeks
  Predialysis serum concentration of IL-6 as a measure of inflammation
Change in Stork balance test time | baseline, 8 weeks, 16 weeks
  Stork balance test time as a measure of balance
Change in sit-and-reach test distance | baseline, 8 weeks, 16 weeks
  Sit-and-reach test distance as a measure of flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Buturović Ponikvar, MD, PhD, Study Chair — UMC Ljubljana
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Bogataj S, Pajek J, Buturovic Ponikvar J, Pajek M. Functional training added to intradialytic cycling lowers low-density lipoprotein cholesterol and improves dialysis adequacy: a randomized controlled trial. BMC Nephrol. 2020 Aug 18;21(1):352. doi: 10.1186/s12882-020-02021-2. PMID 32811448